CLINICAL TRIAL: NCT02495792
Title: Using Real Time Biofeedback to Alter Running Biomechanics
Brief Title: Using Real Time Biofeedback to Alter Running Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamie Morris, Physical Therapy Sports Medicine Fellow, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 404239-2
Record Dates: First submitted 2015-05-25; First posted 2015-07-13 (Estimated); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Group does not receive the biofeedback sensor
- Biofeedback group (Experimental): Group does receive the biofeedback sensor
  Interventions: Device: Biofeedback Sensor

INTERVENTIONS:
Device: Biofeedback Sensor — Tibia accelerometer strapped to distal tibia to detect tibial shock
  Arms: Biofeedback group

SUMMARY:
The purposes of this study are 1) to assess foot strike patterns initially, at six months and at one year between two groups of runners attempting to transition to a non-rearfoot strike pattern (NRFS) with and without the use of biofeedback technology, and 2) to prospectively compare injury incidence rates at one year between NRFS and rearfoot strike (RFS) runners.

ELIGIBILITY:
Inclusion Criteria:

1. Between the age of 18 - 50 years
2. Run on average 12mi per week
3. DOD beneficiaries who intend to remain at West Point, NY for the next 12 months at time of study enrollment
4. Read and speak English well enough to provide informed consent and follow study instructions

Exclusion Criteria:

1. Known pregnancy currently or in the previous 6 months
2. Lower extremity or low back pain in the previous 3 months
3. Lower extremity or low back surgery in the previous 6 months
4. Any lower extremity or low back exercise limiting profile
5. Previous stress fracture of the foot
6. Participant who has a non-rearfoot strike running pattern

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 191 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie B Morris, DPT, Principal Investigator — Keller Army Community Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Biofeedback Group
Started | 96 | 95
Completed | 59 | 55
Not Completed | 37 | 40
Not completed — Lost to Follow-up | 5 | 9
Not completed — Protocol Violation | 32 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Biofeedback Group | Total
Number analyzed (Participants) | 59 | 55 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (9.6) | 25.7 (9.1) | 26.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 44 | 44 | 88
Height [Mean (Standard Deviation); unit: Centimeters] | 173.1 (12.2) | 174.9 (8.3) | 174 (10.2)
Weight [Mean (Standard Deviation); unit: Kilograms] | 74.3 (12.4) | 75.8 (11.8) | 75.1 (12.1)
Weekly Mileage [Mean (Standard Deviation); unit: Kilometers per Week] | 23.7 (10.7) | 22.9 (14) | 23.3 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Foot Strike Pattern From Baseline
Description: Foot strike pattern will be either classified as rearfoot strike or non-rearfoot strike. This is determined by video analysis of 240hz camera. All participants baseline foot strike pattern was rearfoot at study enrollment.
Time Frame: Immediately post-training, 6mo post-training, and 1yr post-training
Measure: Number; unit: percentage of non-rearfoot strike patter
Arm/Group | Control Group | Biofeedback Group
Number analyzed (Participants) | 59 | 55
percentage of non-rearfoot strike patter
  Post-Training | 79 | 83
  6 months | 68 | 73
  1 year | 69 | 75

2. Secondary Outcome: Injury Incidence Between Foot Strike Patterns
Description: Percentage of runners that became injured over 1 yr. Injury defined as pain in the lower extremity that caused restriction or stoppage of running for at least one week, or required the runner to consult a physician or other health care professional.
Time Frame: 1yr
Measure: Number; unit: percentage of injured runners
Groups:
- Rearfoot Strike Pattern: Runners that have initial foot contact as rearfoot strike
- Non-rearfoot Strike Pattern: Runners with an initial foot contact of non-rearfoot strike
Arm/Group | Rearfoot Strike Pattern | Non-rearfoot Strike Pattern
Number analyzed (Participants) | 32 | 82
percentage of injured runners | 37 | 30

3. Secondary Outcome: Relative Risk of Injury
Description: Risk of runner to develop a knee injury based on foot-strike pattern
Time Frame: 1yr
Measure: Count of Participants; unit: Participants
Groups:
- Rearfoot Strike Pattern (RFS): Runners that have initial foot contact as rearfoot strike
- Non-rearfoot Strike Pattern (NRFS): Runners with an initial foot contact of non-rearfoot strike
Arm/Group | Rearfoot Strike Pattern (RFS) | Non-rearfoot Strike Pattern (NRFS)
Number analyzed (Participants) | 32 | 82
Participants
  Developed knee pain | 7 | 3
  Did not develop knee pain | 25 | 79
Statistical Analysis 1: Comparison: Rearfoot Strike Pattern (RFS); Test type: Other; Risk Ratio (RR) = 5.98, 95% CI 2-sided [1.6 to 21.7]

ADVERSE EVENTS:
Arm/Group | Control Group | Biofeedback Group
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/95
Other Adverse Events (participants affected / at risk) | 0/96 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No